CLINICAL TRIAL: NCT05519475
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of siRNA Gene Silencing for the Treatment of Metabolic Dysfunction-Associated Steatohepatitis (MASH) in Participants With Genetic Risk Factors
Brief Title: A Precision Medicine Approach Using Gene Silencing to Treat a Chronic Liver Disease Called Metabolic Dysfunction-Associated Steatohepatitis (MASH) in Adult Participants at Increased Genetic Risk for This Condition
Acronym: NASHGEN-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-HSD-NASH-2130
Record Dates: First submitted 2022-08-15; First posted 2022-08-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction-associated Steatohepatitis (MASH)
Keywords: Metabolic dysfunction-associated steatotic liver disease (MASLD); Histologically confirmed MASH; Genetic risk alleles for MASH at the HSD17B13 locus; Non-alcoholic steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALN-HSD (Experimental): Randomized 1:1
  Interventions: Drug: ALN-HSD
- Placebo (Placebo Comparator): Randomized 1:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-HSD — Administered by subcutaneous injection (SC)
  Arms: ALN-HSD
Drug: Placebo — Administered by SC injection
  Arms: Placebo

SUMMARY:
This study is researching an investigational drug, ALN-HSD called "study drug". This study is focused on participants who are known to have metabolic dysfunction-associated steatohepatitis (MASH). MASH is a form of metabolic dysfunction-associated steatotic liver disease (MASLD). MASH occurs when fat builds up in liver cells, damaging them, and making the liver inflamed and stiff from fibrosis (scar tissue). MASH can progress to cirrhosis (long term scarring) and liver failure (when the liver cannot perform its job). The aim of the study is to see the effect of the study drug on lessening liver scarring side effects related to MASH.

The study is looking at several other research questions, including:

* How ALN-HSD works to improve liver function and lessen MASH-related inflammation in the liver
* What side effects may happen from receiving the study drug
* How much study drug and study drug metabolites (byproduct of the body breaking down the study drug) are in the blood at different times
* Better understanding of the study drug and MASH

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult male or female ≥18 years (or country's legal age of adulthood)
2. A diagnosis of MASH with fibrosis (F) stage 2 or 3, according to the NASH-Clinical Research Network (CRN)
3. NAS score ≥3, as defined in the protocol
4. Meets genotype criteria for study enrollment, as defined in the protocol
5. Has protocol defined FibroScan®-AST (FAST) score at screening or within approximately 12 weeks of screening

Key Exclusion Criteria:

1. Evidence of other forms of known chronic liver disease, as defined in the protocol
2. Known history of alcohol or other substance abuse within the last year or at any time during screening, as defined in the protocol
3. History of Type 1 diabetes
4. Bariatric surgery within approximately 5 years prior to or planned during the study period
5. Prior exposure to any investigational drug targeting HSD17B13 or patatin-like phospholipase domain containing 3 (PNPLA3) (eg, ALN-HSD, ARO-HSD, ALN-PNP, AZD2693)

Note: Other protocol-defined Inclusion/Exclusion Criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2027-09-08 (Estimated); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
Change in qFibrosis | Baseline to week 52
  Change in the continuous quantitative liver fibrosis (qFibrosis) score measured by second harmonic generation/two-photon excitation microscopy

SECONDARY OUTCOMES:
Improvement of non-alcoholic steatohepatitis clinical research network (NASH-CRN) fibrosis (F) stage by ≥1 stage without worsening of MASH on liver biopsy | Baseline to week 52
Resolution of MASH with no worsening of NASH-CRN fibrosis on liver biopsy | Baseline to week 52
  Resolution of MASH (steatohepatitis) is defined as absent fatty liver disease or isolated or simple steatosis without steatohepatitis and a non-alcoholic fatty liver disease activity score (NAS) score of 0-1 for inflammation, 0 for ballooning, and any value for steatosis
Change in serum alanine aminotransferase (ALT) | Baseline to week 52
Change in serum aspartate aminotransferase (AST) | Baseline to week 52
Change in enhanced liver fibrosis (ELF) | Baseline to week 52
Change in N-terminal type III collagen propeptide (PRO-C3) | Baseline to week 52
Change in NIS4, a non-invasive fibrosis biomarker of NASH | Baseline to week 52
Change in Fibrosis-4 (FIB-4) | Baseline to week 52
Change in hepatic hydroxysteroid 17β dehydrogenase 13 (HSD17B13) transcript level | Baseline to week 52
Incidence of progression in qFibrosis on liver biopsy | Baseline to week 52
Incidence of treatment-emergent adverse events (TEAEs) | Baseline to week 84
Severity of treatment-emergent adverse events (TEAEs) | Baseline to week 84

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (71):
- United States (61):
  - Arizona Liver Health, Chandler, Arizona
  - The Institute for Liver Health II LLC DBA Arizona Clinical Trials - Flagstaff, Flagstaff, Arizona
  - The Institute for Liver Health II LLC DBA Arizona Liver Health - Peoria, Peoria, Arizona
  - Adobe Clinical Research, Tucson, Arizona
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - Velocity Clinical Research, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - Velocity Clinical Research, Gardena, California
  - Velocity Clinical Research - Huntington Park, Huntington Park, California
  - Om Research Llc, Lancaster, California
  - Ark Clinical Research - Long Beach, Long Beach, California
  - Velocity Clinical Research - Westlake, Los Angeles, California
  - Clinnova Research Solutions, Orange, California
  - Knowledge Research Center, St. Joseph's Medical Tower, Orange, California
  - National Research Institute, Panorama City, California
  - California Liver Research Institute, Pasadena, California
  - Cadena Care Inst., Poway, California
  - Inland Empire Liver Foundation, Rialto, California
  - Precision Research Institute - San Diego, San Diego, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Synergy Healthcare LLC, Bradenton, Florida
  - Evolution Clinical Trials, Hialeah Gardens, Florida
  - Health Awareness, inc., Jupiter, Florida
  - Miami Clinical Research, Miami, Florida
  - International Medical Investigational Centers (IMIC) Incorporated, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - US Associates in Research, LLC, Miami, Florida
  - Med Research of Florida, LLC, Miami, Florida
  - Charter Research LLC - Orlando, Orlando, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Deaconess Clinic - GI Specialty Center, Newburgh, Indiana
  - Tandem Clinical Research, Metairie, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - GI Associates, Flowood, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Austin Clinical Research, LLC, Austin, Texas
  - American Research Corporation, Austin, Texas
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - South Texas Research Institute (STRI) - Brownsville, Brownsville, Texas
  - Velocity Clinical Research - Austin, Cedar Park, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - South Texas Research Institute (STRI) - Edinburg, Edinburg, Texas
  - GI Alliance Research, Fort Worth, Texas
  - Allure Health at Mt. Olympus Medical Research, Friendswood, Texas
  - Advanced Medical Trials, Georgetown, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - R & H Clinical Research, Inc., Katy, Texas
  - Great Lakes Research Institute, Pharr, Texas
  - American Research Corporation at The Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - R & H Clinical Research, Stafford, Texas
  - Intermountain Health, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Richmond Veterans Administration Medical Center, Richmond, Virginia
- JCHO Hokkaido Hospital, Sapporo, Hokkaido, Japan
- Puerto Rico (4):
  - Isis Clinical Research Center, Guaynabo, San Juan
  - Klinical Investigations, San Juan
  - Latin Clinical Trial Center, San Juan
  - Fundacion de Investigacion (FDI) Clinical Research, San Juan
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Hanyang University Seoul Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * has the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Study Informational Website — https://nashgenstudy.com/en-us